CLINICAL TRIAL: NCT04115046
Title: Pilot Study Evaluating Endoscopic Ultrasound With ShearWave Elastography for Diagnosis and Staging of Liver Fibrosis
Brief Title: The EUS ShearWave Elastography Liver Fibrosis Study
Status: Completed | Type: Observational
Sponsor: Olympus Corporation of the Americas (Industry)
Collaborators: Geisinger Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-GI-ShearWave
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Liver Fibroses
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment Arm: Consecutive, eligible patients reporting for an ultrasound and liver biopsy for evaluation of fibrosis will be enrolled. Each subject will undergo both procedures (FibroScan and EUS with SW Elastography).
  Interventions: Device: ShearWave Elastography (SWE) in Endoscopic Ultrasound (EUS); Device: FibroScan; Device: ALOKA ARIETTA 850 -

INTERVENTIONS:
Device: ShearWave Elastography (SWE) in Endoscopic Ultrasound (EUS) — ShearWave Measurement is a software option available on the ARIETTA 850 that uses transient pulses to generate shear waves in the body. The tissue's elasticity is directly deduced by measuring the speed of wave propagation.
Device: FibroScan — manufactured by Echosens
Device: ALOKA ARIETTA 850 - — manufactured by Hitachi Healthcare - included on the system is the ShearWave measurement software

SUMMARY:
The study objective is to demonstrate the clinical performance of ShearWave Elastography (SWE) in Endoscopic Ultrasound (EUS) when compared to FibroScan for evaluation of liver fibrosis.

DETAILED DESCRIPTION:
This study has been designed as prospective, single center, single arm, consecutive, blinded, pilot study conducted in a post-market setting using commercially available devices to evaluate the effectiveness of Endoscopic Ultrasound with ShearWave Elastography to estimate hepatic fibrosis in patients with chronic liver disease. It is anticipated that the data from this study will support the need for additional clinical trials. All consenting, eligible patients reporting for an ultrasound and/or liver biopsy for evaluation of fibrosis meeting the inclusion criteria will be consecutively enrolled into the study and assigned a unique study identification number. A total of 52 subjects will be enrolled and treated at a single study site in the US. Enrollment is expected to be completed within 6 months. Each subject will undergo both procedures (FibroScan and EUS with SW Elastography), End of study will be reached after pathology results have been obtained (within a week of the initial procedure).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Willing and able to provide informed consent
3. Undergoing diagnostic EUS procedure with liver biopsy
4. Baseline CBC, CMP, INR within 3 months

Exclusion Criteria:

1. Contraindication to EUS-guided liver biopsy
2. Baseline platelet count <50,000
3. Baseline INR >1.5
4. Patient is a prisoner

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consenting, eligible patients reporting for an ultrasound and/or liver biopsy for evaluation of fibrosis.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Analyze the correlation between SWE of liver and FibroScan of liver with histologic fibrosis stage using Spearman Correlation Coefficient. | 6 months
  Use ANOVA with Tukey Range test to evaluate the level of significance of difference in SWE results across fibrosis stages.
Analyze the correlation between SWE of liver and FibroScan of liver with histologic fibrosis stage using Spearman Correlation Coefficient. | 6 months
  Construct receiver operating characteristic curves (ROC) to determine which liver section (left or right) had best accuracy of prediction of fibrosis stage and compared overall accuracy between SWE and TE.

CONTACTS AND LOCATIONS:
Overall Officials: David Diehl, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be accessible starting 6 months after publication

REFERENCES:
- [Derived] Termite F, Borrelli de Andreis F, Liguori A, Gasbarrini A, Attili F, Spada C, Miele L. The Role of Endoscopic Ultrasound in Assessing Portal Hypertension: A State-of-the-Art Literature Review and Evolving Perspectives. Liver Int. 2025 Apr;45(4):e16176. doi: 10.1111/liv.16176. Epub 2024 Nov 27. PMID 39601324